CLINICAL TRIAL: NCT06947161
Title: The Pilot Study of Throat Packs Soaked in Gengigel Spray in Patients Undergoing Elective Surgery Under General Anaesthesia
Brief Title: Pilot Study of Throat Packs Soaked in Gengigel Spray in Patients Undergoing Elective Surgery
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, SABREENA BINTI ISMAIL, Principal Investigator, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024917-14215
Record Dates: First submitted 2025-04-02; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Throat, Sore
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Intervention Model Description: rct
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline soaked throat pack (Experimental): Throat pack used will be soaked with saline
  Interventions: Drug: Gengigel
- Gengigel soaked throat pack (Experimental): Throat pack used will be soaked with gengigel
  Interventions: Drug: Gengigel

INTERVENTIONS:
Drug: Gengigel — Throat pack will be soaked with gengigel, and post operatively, will see if there is any presence of sore throat, severity of sore throat. 10 mlm of gengigel, in liquid form will be used to soak the throat pack. 30 patients will receive gengigel spray soaked throat pack, and control group will receive normal saline soaked throat pack

SUMMARY:
Throat packs are commonly used in many surgical procedures involving the oral cavity and pharynx, primarily to prevent blood, saliva, and other debris from entering the lower respiratory tract, thereby maintaining a clear airway and reducing the risk of aspiration and respiratory complications. Traditionally, these packs are moistened with saline or used in a dry state, with the choice often depending on the surgeon's preference and specific surgical requirements. However, despite their widespread usage, the exploration of alternative substances to moisten throat packs, particularly those with additional therapeutic benefits, remains limited in medical research. This pilot study introduces Gengigel spray as an innovative alternative to saline for moistening throat packs. Gengigel, a hyaluronic acid (HA)-based product, is known for its healing properties and anti-inflammatory effects, which are beneficial in oral care. Gengigel provides a non-anesthetic approach that promotes tissue repair and reduces inflammation. This makes it particularly advantageous in the context of surgical procedures where reducing postoperative inflammation and promoting mucosal healing are crucial.

DETAILED DESCRIPTION:
Using throat packs is a standard practice in surgeries involving the oral cavity, pharynx, and upper airway to prevent the aspiration of blood and other debris, which could lead to postoperative complications such as aspiration pneumonia. Traditionally, these throat packs are moistened with saline or left dry. However, this conventional approach has been associated with postoperative throat pain and discomfort, which are common and often distressing complications for patients undergoing surgery under general anesthesia. The discomfort caused by these packs can delay recovery, extend hospital stays, and negatively impact overall patient satisfaction with the surgical experience.

Gengigel presents a novel alternative with distinct advantages. Gengigel, which contains hyaluronic acid (HA), is recognized for its anti-inflammatory and healing properties, making it a promising candidate for improving postoperative outcomes when used in throat packs. Despite Gengigel's established use in other medical applications, such as wound care and oral health, there is currently no research exploring its effectiveness in moistening throat packs during surgical procedures. This represents a significant knowledge gap, as the combination of Gengigel's healing and anti-inflammatory effects could potentially address both pain and mucosal recovery.

Addressing this gap is crucial for advancing postoperative care, as current literature does not adequately explore the potential benefits or risks associated with using Gengigel in throat packs. Furthermore, there is a lack of data on patient outcomes, including the extent of pain relief, the speed of mucosal healing, potential complications, and overall patient satisfaction when Gengigel is utilized in this context. The absence of such data limits the ability of healthcare providers to make evidence-based decisions that could improve patient care.

To bridge this gap, this study proposes a randomized controlled trial (RCT) to compare the outcomes of using Gengigel-soaked throat packs versus traditional saline-soaked packs in patients undergoing surgery under general anesthesia. The study will systematically assess postoperative throat pain levels, evaluate the degree of mucosal healing, monitor for any adverse effects, and measure overall patient satisfaction. By conducting this comprehensive evaluation, the research aims to provide robust evidence that could guide the use of Gengigel in throat packs, potentially setting a new standard in postoperative care. Ultimately, the findings could lead to enhanced patient comfort, faster recovery times, and a higher quality of care for patients undergoing surgeries involving the oral cavity and pharynx.

ELIGIBILITY:
Inclusion Criteria:

1. Classified as ASA I-II, indicating a relatively low risk of complications from anesthesia
2. Aged between 18 and 60 years, which represents a typical adult surgical population
3. Both male and female patients, ensuring gender inclusivity and representation in the study findings

Exclusion Criteria:

1. Existing sore throat prior to surgery, which could affect the baseline measurement of postoperative sore throat.
2. Anticipation of a difficult airway, as these patients may require specialized intubation techniques that are not standardized across the study.
3. More than two attempts at endotracheal tube (ETT) insertion, as multiple attempts could cause additional trauma and skew the study outcomes.
4. Any trauma occurring during intubation, which could independently contribute to postoperative sore throat and other complications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-08-12 (Estimated); Study Completion 2025-08-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative sore throat. | 6 months
  This will be assessed with Scoring System of Harding and McVey

SECONDARY OUTCOMES:
Severity of postoperative sore throat | 6 months
  This will be assessed with Scoring System of Harding and McVey
Patient satisfaction | 6 months
  This will be assessed with a yes/no question regarding their overall satisfaction with the postoperative care.
The presence of hoarseness of voice | 6 months
  This will be assessed with Scoring System of Harding and McVey
The presence of cough | 6 months
  This will be assessed with Scoring System of Harding and McVey

CONTACTS AND LOCATIONS:
Locations (1):
- Sabreena Ismail, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-16): https://cdn.clinicaltrials.gov/large-docs/61/NCT06947161/Prot_SAP_000.pdf